CLINICAL TRIAL: NCT05612217
Title: A Study to Evaluate a Accuracy of the AIVARIX AI-based Application in Detecting Signs C 1-2 Classes of CVD in Outpatients Seeking Consultancy of Phlebologists in the Russian Federation
Brief Title: Evaluation of the AIVARIX in Detecting Signs C 1-2 Classes of CVD
Acronym: AIVARIX
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-05682-071-RUS
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Chronic Venous Disease; CVD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with CVD: 20 patients per 1 center: patients with CVD C1 class 4 patients with CVD C2 class; 2 patients with CVD with classes other than C1-C2 (C4-C6); 8 patients with either C0s CVD or with skin pathologic conditions of lower extremities other than CVD;
  Interventions: Other: to estimate Sensitivity and Specificity AIVARIX app in detecting C1 and C2 classes of CVD

INTERVENTIONS:
Other: to estimate Sensitivity and Specificity AIVARIX app in detecting C1 and C2 classes of CVD — to estimate Sensitivity and Specificity of the AI-based AIVARIX app in detecting C1 and C2 classes of CVD in patients who are seeking for professional advice from a phlebologist regarding symptoms and signs suggestive to CVD.

SUMMARY:
This study is a multicenter observational study, which is carried out in frame of routine clinical practice in Russia. The program will include patients suggestive to chronic venous diseases (CVDs) including but not limited to those with C1 and C2 classes by CEAP classification, who will be seeking professional phlebologists' consultation. Study conduction is scheduled in Russia in 2022-2023. The planned number of patients is 414

DETAILED DESCRIPTION:
The main goal of this study is to describe the AIVARIX app accuracy in detecting C1 and C2 classes by CEAP classification of chronic venous disease (CVD) in patients who are consulted by phlebologists on symptoms and signs suggestive to CVD.

At single visit, investigating physicians (phlebologists) will be assessing and collecting parameters of interest which they should input in eCRF.

Following data will be collected at the visit: a signed consent form from a patient, demographic characteristics (age, sex), eligibility of a patient to the inclusion/ non-inclusion criteria, 1 (one) image of skin area of interest, conclusion on presence or absence of CVD or any other pathologic condition(s) made as a result of objective/ instrumental examination. In case there will be any information related to safety of a Servier drug provided, investigating physician will also collect the information and fill in the PV form (Appendix 1).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Written informed consent is provided
* Symptoms and signs of CVD or any other skin pathologic condition (s) of lower extremities for which a patient seeks for phlebologist's consultation
* Ability to fulfil the technical requirements for smartphones/ images

Exclusion Criteria:

* Patients with mental/ psychiatric disabilities who are not able to understand objectives of the study and therefore provide a signed consent to participate in the study.
* Patient's decision to withdraw his/her consent to participate in the study at any moment of the study conduction

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who are consulted by phlebologists on symptoms and signs suggestive to CVD.
Sampling Method: Non-Probability Sample
Enrollment: 433 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: IGOR ZOLOTUKHIN, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- Pirogov Russian National Research Medical University, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With CVD
Started | 433
Completed | 433
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With CVD
Number analyzed (Participants) | 433
Age, Continuous [Median (Standard Deviation); unit: years] | 46 (18.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 332
  Male | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 433

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Sensitivity (Sn) of the AI-based AIVARIX App in Detecting C1 and C2 Classes of CVD in Patients Who Are Seeking for Professional Advice From a Phlebologist Regarding Symptoms and Signs Suggestive to CVD.
Description: Sensitivity is defined as the ratio of the number of positive cases of detection of signs of C1 or C2 CVD, identified using the AIVARIX tool, to the total number of truly positive cases of C1 or C2 CVD in the study population, confirmed by phlebologists using objective / instrumental examinations.
Time Frame: 1 month
Measure: Number (95% Confidence Interval); unit: percentage of of positive cases
Arm/Group | Patients With CVD
Number analyzed (Participants) | 433
percentage of of positive cases | 75.19 [66.82 to 82.37]

2. Primary Outcome: Evaluation of Specificity (Sp) of the AI-based AIVARIX App in Detecting C1 and C2 Classes of CVD in Patients Who Are Seeking for Professional Advice From a Phlebologist Regarding Symptoms and Signs Suggestive to CVD
Description: Specificity is defined as a proportion of the number of negative cases of signs C1 or C2 classes of CVD identified by the AIVARIX tool divided to overall truly negative cases of C1 or C2 in the study population confirmed by phlebologists by means of objective/ instrumental examination.
Time Frame: 1 month
Measure: Number (95% Confidence Interval); unit: percentage of negative cases
Arm/Group | Patients With CVD
Number analyzed (Participants) | 433
percentage of negative cases | 86.51 [82.15 to 90.14]

3. Secondary Outcome: Calculation of the Positive Predictive Values (PPV) a of AIVARIX in Detecting Signs of C1 and C2 Classes of Chronic Venous Disease.
Description: PPV is defined as the proportion of true positive cases of class C1 or C2 CVD detected using AIVARIX as a proportion of the number of true positive and false positive cases of class C 1 or C 2 identified using the AIVARIX application and confirmed by phlebologists.
Time Frame: 1 month
Measure: Number (95% Confidence Interval); unit: percent of positive predictive values
Arm/Group | Patients With CVD
Number analyzed (Participants) | 433
percent of positive predictive values | 70.29 [61.92 to 77.76]

4. Secondary Outcome: Calculation of the Negative Predictive Values (NPV) a of AIVARIX in Detecting Signs of C1 and C2 Classes of Chronic Venous Disease.
Description: The NPV is defined as the ratio of the number of true negative cases of C 1 or C 2 CVD detected using AIVARIX to the true negative and false negative cases of C 1 or C 2 CVD detected using AIVARIX and confirmed by phlebologists.
Time Frame: 1 month
Measure: Number (95% Confidence Interval); unit: percentage of negative predictive values
Arm/Group | Patients With CVD
Number analyzed (Participants) | 433
percentage of negative predictive values | 89.15 [85.03 to 92.46]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Patients With CVD
All-Cause Mortality (participants affected / at risk) | 0/433
Serious Adverse Events (participants affected / at risk) | 0/433
Other Adverse Events (participants affected / at risk) | 0/433

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT05612217/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT05612217/ICF_001.pdf